CLINICAL TRIAL: NCT03589625
Title: Evaluation of the Impact of the 'Solar Suitcase' Installation in Healthcare Facilities in Uganda on Quality of Care During Labor and Delivery and Reliability of Electricity
Brief Title: Electricity Access and Maternal Care in Rural Health Facilities in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: University College Dublin (Other); Innovations for Poverty Action (Other)
Responsible Party: Principal Investigator, Jessica Cohen, Associate Professor of Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-18-0406
Record Dates: First submitted 2018-06-07; First posted 2018-07-18 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Quality of Care
Keywords: electricity and health; maternal health; quality of care; solar power

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solar Suitcase Installation First Group (Experimental): Facilities will receive the installation of the Solar Suitcase shortly after baseline data collection.
  Interventions: Other: Solar Suitcase
- Solar Suitcase Installation Second Group (Experimental): Facilities will act as a comparator for experimental group 1 and then will receive the installation of the Solar Suitcase shortly after midline data collection.
  Interventions: Other: Solar Suitcase

INTERVENTIONS:
Other: Solar Suitcase — The intervention is a "Solar Suitcase". The Solar Suitcase comes with: 2 LED lights, 1 battery, 1 aluminum glass 100 watt solar panel, 2 rechargeable LED headlamps, 1 universal cell phone charger, 1 USB adapter, 1 fetal Doppler, 1 AA/AAA battery charger and expansion box (provides 2 additional lights).
  Installers will teach health workers how to use and maintain the Solar Suitcase on the day of installation. Within one week following installation, the contractor will contact the facility over the phone and/or in-person to check if there are any problems with the Suitcase. Additional checks will be made to ensure the solar suitcase is functioning and being used properly.

SUMMARY:
The investigators will conduct a stepped wedge cluster-randomized controlled trial in maternity care facilities in Uganda to evaluate the impact of the provision of a reliable light source on the quality of delivery care provided. The facility-level intervention is the installation of a "Solar Suitcase", a complete solar electric system providing essential lighting and power for charging phones and small medical devices and a fetal doppler. The intervention will be rolled-out sequentially to all facilities over two time periods, in a randomized order.

DETAILED DESCRIPTION:
Ensuring universal access to electricity is essential for global development. In the health sector, lack of reliable light and electricity is a major challenge for health workers when conducting deliveries at night. However, there is very little evidence of the impact of improving access to reliable electrification at maternity facilities on the quality of maternity care they provide.

This stepped wedge cluster-randomized trial will evaluate the impact of a reliable light and electricity source - the "Solar Suitcase" - on outcomes of availability and brightness of light, the quality of maternal care provided, and health worker satisfaction. The study will take place in rural health facilities conducting deliveries in Uganda. The eligible facilities have either no connection to electricity or a modern light source or have reported to have very unreliable light (blackouts occur frequently).

The intervention is a "Solar Suitcase", provided by the non-governmental organization "We Care Solar". The Solar Suitcases are complete solar electric systems that provide essential lighting and power for charging phones and small medical devices. Data collection will include direct observation of deliveries during daytime and nighttime hours, as well as interviews with facility staff. The intervention will be implemented in about 30 facilities in a step process, whereby at each 'step', half of the facilities (selected randomly) will receive the intervention.

Data will be collected at three time points: a baseline period in which no facilities have received the intervention, a midline period in which the first group of facilities has received the intervention but the other half has not, and an endline period in which all facilities have received the intervention.

In addition, facility-level data will be collected at three time points over a 9-month period after the completion of the endline. This data will be used to monitor delivery and ANC volumes at facilities.

ELIGIBILITY:
For women delivering at facility:

Inclusion Criteria:

* Pregnant women who are admitted for labor and delivery at participating facilities.
* Women aged 16 years or older.

Exclusion Criteria:

* Pregnant women who present to participating facilities for abortion or abortion-related complications, miscarriage, ectopic pregnancy, antenatal or postnatal complications of pregnancy (not an observation of labor)
* Women who are immediately transferred to another hospital, or are taken straight to surgical theatre (limited or no period of observation possible)
* Women who deliver at home but are brought to the facility for any complication.
* Women who deliver outside the maternity ward or delivery area
* Women who deliver in ambulance while on the way to the facility (woman admitted in the facility for placenta removal)
* Women who have not given consent
* Health worker objects to the observation.

For eligibility of health facility:

Inclusion criteria:

* government health facilities level 2, 3, or 4
* are open 24 hours a day
* conduct deliveries at night
* have unreliable electricity (have either no source of electricity, or have only 1 functional source of electricity and experience blackouts at least several times a week and had power available only sometimes in the past week).

Exclusion criteria:

• facility already has a Solar Suitcase

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1268 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Average brightness of room during labor and delivery as measured by observer recorded questionnaire | up to 6 months after installation
  Scale is scored as 1: Very Bright; 2: Somewhat Bright; 3: Dim; 4: Pitch Black. Variable is binary indicator for "very bright" or "somewhat bright" throughout delivery
Satisfactory light source used for entire delivery as measured by observer recorded questionnaire | up to 6 months after installation
  Satisfactory light source is a variable equal to 1 if observation occurs without daylight and facility is using grid, solar or functional generator and zero if using kerosene, candle, torch, etc. Variable is always equal to 1 during daylight.
Adequate Light as measured by observer recorded questionnaire | up to 6 months after installation
  Binary variable equal to 1 if light is from a satisfactory source and is "bright" ("very bright" or "somewhat bright") for duration of delivery observation.
20-item quality of maternal care index of essential actions to be performed by provider during labor and delivery as measured by observer recorded questionnaire | up to 6 months after installation
  Quality of care index is based on essential actions providers must perform during the course of labor and delivery, as described in Tripathi et al. (2015). Score is the fraction of 20 items, yielding a range of 0 to 1, with higher scores indicating better quality of maternal care.
37-item quality of maternal care index of essential actions to be performed by provider during labor and delivery as measured by observer recorded questionnaire | up to 6 months after installation
  Quality of care index is based on the essential actions providers must perform during the course of labor and delivery, derived from the Maternal and Child Health Integrated Program (MCHIP). It includes the 20 items from Tripathi et al. (2015) plus an additional 17 quality of care items from MCHIP (2013). Score is fraction of the 37 items, yielding a range of 0 to 1, with higher scores indicating better quality of maternal care.
6-item delays in care index as measured by observer recorded questionnaire | up to 6 months after installation
  Index including:
  i) Time between facility arrival and first contact with health worker (mins) ii) Time between facility arrival and first assessment (mins) iii) Time between delivery and uterotonic (mins) iv) Time between delivery and assessment of perineal and vaginal lacerations (mins) v) Time between delivery and drying baby with towel (mins) vi) Time between delivery and initiation of breastfeeding (mins) Score is average of the 6 items measured in minutes, with lower values indicating reduced delays in quality of maternal care. Range from 0 to 120 minutes.
Health Worker Satisfaction with Electricity as measured by health worker survey | up to 6 months after installation
  Responses on a 1-5 scale with 1: Strongly Disagree, 2: Disagree, 3: Neutral (Neither Agree nor Disagree), 4: Agree, 5: Strongly Agree
  Worker Satisfaction with Electricity is a binary variable equal to 1 if strongly agree with both:
  i) I am satisfied with the availability and brightness of light in this facility.
  ii) I am satisfied with the availability of electricity in this facility
Overall job satisfaction index as measured by health worker survey | up to 6 months after installation
  Responses on a 1-5 scale with 1: Strongly Disagree, 2: Disagree, 3: Neutral (Neither Agree nor Disagree), 4: Agree, 5: Strongly Agree
  Overall job satisfaction index is the mean score (1-5) of the 4 below components:
  i) These days, I feel motivated to work as hard as I can. ii) Overall, I am satisfied with my job. iii) Overall, the morale level at my department is good iv) I plan on staying at this position for the next year.

SECONDARY OUTCOMES:
Mean level of brightness over 4 periods of labor and delivery on brightness scale as measured by observer recorded questionnaire | up to 6 months after installation
  Scale is scored as 1: Very Bright; 2: Somewhat Bright; 3: Dim; 4: Pitch Black
Minutes of delivery observation without satisfactory light as measured by observer recorded questionnaire | up to 6 months after installation
  Satisfactory light source defined in Primary Outcome 2.
Consistent satisfactory light source as measured by observer recorded questionnaire | up to 6 months after installation
  Variable equal to 1 if no interruptions of > 2 hours in satisfactory light source during observed deliveries.
Fetal Doppler Use as measured by observer recorded questionnaire | up to 6 months after installation
  Number of times the provider used a fetal doppler during labor and delivery
Phone availability as measured by observer recorded questionnaire | up to 6 months after installation
  Phone is available and on for deliveries
APGAR Score Assigned as measured by observer recorded questionnaire | up to 6 months after installation
  Provider assigns any APGAR score (binary variable equal to 1 if provider assigns an APGAR score (range of 0-10), and equal to 0 if no APGAR score is assigned.
Basic emergency obstetric care signal functions as measured by facility assessment | up to 6 months after installation
  Facility reported performance of basic emergency obstetric care signal functions in the past three months. Measure includes the number of signal functions performed from:
  1. Removal of retained products of conception
  2. Parenteral oxytocin for maternal hemorrhage
  3. Parenteral magnesium sulfate for (pre-) eclampsia
  4. Manual removal of placenta
  5. Parenteral antibiotics for maternal infection
  6. Assisted vaginal delivery
Basic emergency newborn care signal functions as measured by facility assessment | up to 6 months after installation
  Facility reported performance of basic emergency newborn care signal functions in the past three months. Measure includes the number of signal functions performed from:
  1. Antibiotics for preterm or prolonged PROM
  2. Corticosteroids in preterm labor
  3. Resuscitation with bag and mask for non-breathing baby
  4. Kangaroo Mother Care for premature/very small babies
  5. Alternative feeding if baby unable to breastfeed
  6. Injectable antibiotics for neonatal sepsis
  7. PMTCT if HIV-positive mother
Routine obstetric care signal functions as measured by facility assessment | up to 6 months after installation
  Facility reported universal practice of routine obstetric care signal functions. Measure includes the number of signal functions performed from:
  1. Infection control (provider hand-washing before patient exam in labor, new sterile gloves before every vaginal examination)
  2. Use of partograph to monitor labor
  3. Routine practice of active management of the third stage of labor
Routine newborn care signal functions as measured by facility assessment | up to 6 months after installation
  Facility reported universal practice of routine newborn care signal functions. Measure includes the number of signal functions performed from:
  1. Thermal protection (newborn dried immediately, skin-to-skin, no bath/delayed>6 hours)
  2. Exclusive breastfeeding initiated within 1 hour of birth
  3. Hygienic cord care (cord cut with sterile blade/scissors; chlorhexidine or nothing applied to stump)
Time between delivery and when suturing began (minutes) as measured by observer recorded questionnaire | up to 6 months after installation
  Observed time between delivery and when provider began suturing lacerations, if needed.
4-item quality of suturing index as measured by observer recorded questionnaire | up to 6 months after installation
  Index constructed from the following variables:
  * Health worker explains to woman what is happening (binary)
  * Health worker cleans area prior to suturing with antiseptic solution (binary)
  * Health worker prepares instruments/sutures on a sterile surface (binary)
  * Health worker sutures episiotomy or tears appropriately in layers. (binary) Score is fraction of 4 items, yielding a range of 0-1, with higher score indicating better quality of suturing.
10-item patient treatment index as measured by observer recorded questionnaire | up to 6 months after installation
  Patient treatment/inter-personal quality care index, based on Kruk et al. (2014) including whether health worker: shouted/scolded patient, threatened to withhold treatment, ignored/left patient, did not answer questions, was not present when delivery began, slapped/beat mother, stitched episiotomy without anesthesia, demanded payment inappropriately, requested bribe, did not provide privacy to mother. Fraction of items that were NOT performed, yielding a range of 0-1, with higher scores indicating better treatment of patients.
14-item Partograph Completeness index as measured by observer recorded questionnaire | up to 6 months after installation
  Index of variables (from MCHIP (2013) tool capturing completeness of recording on partograph). Fraction of 14 items completed on partograph (all binary variables), yielding a range of 0-1, with higher values indicating more completeness.
Time between contractions as measured by observer recorded questionnaire | up to 6 months after installation
  Time between contractions at first exam (mins)
Dilation at first exam as measured by observer recorded questionnaire | up to 6 months after installation
  Degree of dilation at woman's first exam (cm)
Monthly Delivery Volumes as measured by facility register | up to 6 months after installation
  Average Number of Monthly Deliveries
Monthly Nighttime Delivery Volumes as measured by facility register | up to 6 months after installation
  Average Number of Nighttime Deliveries per Month
Monthly ANC Volumes as measured by facility register | up to 6 months after installation
  Average Number of Antenatal Clients per Month
Monthly Referral Volumes as measured by facility register | up to 6 months after installation
  Average Number of Monthly Referrals Out of Facility for Mothers and Newborns
Sensor Brightness as measured by sensor | up to 6 months after installation
  Recorded brightness at sensor sight in the two hours around delivery of baby.
Depletion of Solar Suitcase Battery Based on Voltage as measured by sensor | up to 6 months after installation
  Average difference between solar suitcase load voltage in evening and morning (based on sensor)
Depletion of Solar Suitcase Battery Based on Charge Time as measured by sensor | up to 6 months after installation
  Average time between morning and when the solar suitcase is fully charged, based on sensor
Solar Suitcase Use for Deliveries as measured by enumerator recorded questionnaire | up to 6 months after installation
  Fraction of deliveries in which enumerator recorded usage of suitcase
Health Worker Assessment of Overhead Light Availability as measured by health worker survey | up to 6 months after installation
  Health worker response (1-5) on the following scale: 1: No overhead light; 2: Very poor; 3: Poor; 4: Good; 5: Very Good to the question:
  "In general, how would you rate the availability of overhead light for maternal and newborn care (deliveries) in this facility at night?"
Health Worker Assessment of Task Light Availability as measured by health worker survey | up to 6 months after installation
  Health worker response (1-5) on the following scale: 1: No procedure/task light; 2: Very poor; 3: Poor; 4: Good; 5: Very Good to the question:
  "In general, how would you rate the availability of procedure/task light for maternal and newborn care (deliveries) in this facility at night?"
Health Worker Assessment of Overhead Light Brightness as measured by health worker survey | up to 6 months after installation
  Health worker response (1-5) on the following scale: 1: No overhead light; 2: Very poor; 3: Poor; 4: Good; 5: Very Good to the question: "In general, when the overhead light is on, how would you rate the quality of light (brightness) for maternal and newborn care (deliveries) in this facility at night?"
Health Worker Assessment of Task Light Brightness as measured by health worker survey | up to 6 months after installation
  Health worker response (1-5) on the following scale: 1: No procedure/task light; 2: Very poor; 3: Poor; 4: Good; 5: Very Good to the question: "In general, when the procedure/task light is on, how would you rate the quality of light (brightness) for maternal and newborn care (deliveries) in this facility at night?"
14-item index of Health worker assessment of impact of blackouts on their ability to perform job functions as measured by health worker survey | up to 6 months after installation
  Index of items measuring health worker assessment of impact of blackouts in facility on ability to conduct their job, including how often health worker: conducted deliveries without overhead light; had to hold torch in hand to see patient; experienced lack of light that affected normal care provided; delayed care; feared to move around facility; was affected in ability to suture, find/use equipment, conduct examinations of mother, provide emergency care, provide newborn care, monitor fetal heartrate, administer medication, clean up after delivery, manage infection control. Response to items scored (1-5) on following scale: 1. Every delivery, 2. Most, 3. Some, 4. Few, or 5. Never. Overall score measured as average of 14 items, yielding a range of 1-5.
Initial exam Bleeding Assessment as measured by observer recorded questionnaire | up to 6 months after installation
  Provider asks whether woman has experienced vaginal bleeding during current pregnancy (binary)
Initial exam Headaches/Blurred Vision Assessment as measured by observer recorded questionnaire | up to 6 months after installation
  Provider asks whether woman has experienced headaches and/or blurred vision during current pregnancy (binary)
HIV testing as measured by observer recorded questionnaire | up to 6 months after installation
  Provider offers woman an HIV test or checks her HIV status (binary)
Takes Pulse as measured by observer recorded questionnaire | up to 6 months after installation
  Provider takes pulse of mother during initial exam (binary)
Takes Blood Pressure as measured by observer recorded questionnaire | up to 6 months after installation
  Provider takes both systolic and diastolic blood pressure measurements of mother during initial exam (binary)
Wears Sterile Gloves as measured by observer recorded questionnaire | up to 6 months after installation
  Provider wears sterile gloves for initial vaginal exam (binary)
Communication with Patient as measured by observer recorded questionnaire | up to 6 months after installation
  At least once, explains what will happen in labour to woman and/or her support person. (binary)
Partograph Use as measured by observer recorded questionnaire | up to 6 months after installation
  Provider starts partograph to monitor progress of labour. (binary)
Hand Washing as measured by observer recorded questionnaire | up to 6 months after installation
  Provider washes his/her hands with soap and water or uses alcohol hand rub prior to every examination of woman. (binary)
Preparation of Uterotonic as measured by observer recorded questionnaire | up to 6 months after installation
  Uterotonic is prepared for Active Management of the Third Stage of Labor (AMTSL). (binary)
Preparation of Bag and Mask as measured by observer recorded questionnaire | up to 6 months after installation
  Prepares self-inflating ventilation bag and newborn face mask. (binary)
Administration of Oxytocin as measured by observer recorded questionnaire | up to 6 months after installation
  After delivery, provider administers 10 IU of IM oxytocin, OR:
  * 5 IU slow push if IV in place
  * 600μg of misoprostol sublingually
  * 600μg misoprostol rectally (binary)
Assessment of Completeness of Placenta as measured by observer recorded questionnaire | up to 6 months after installation
  Provider assesses completeness of the placenta and membranes. (binary)
Assessment of Lacerations as measured by observer recorded questionnaire | up to 6 months after installation
  Assesses completeness of the placenta and membranes. (binary)
Skin-to-Skin as measured by observer recorded questionnaire | up to 6 months after installation
  Provider places baby on mother's abdomen or chest skin-to-skin. (binary)
Drying Newborn as measured by observer recorded questionnaire | up to 6 months after installation
  Provider immediately dries baby with towel. (binary)
Cord Clamping as measured by observer recorded questionnaire | up to 6 months after installation
  Provider ties or clamps cord. (binary)
Vital Signs Postpartum as measured by observer recorded questionnaire | up to 6 months after installation
  Provider takes mother's vital signs after delivery. (binary)
Palpation of Uterus as measured by observer recorded questionnaire | up to 6 months after installation
  Provider palpates uterus after delivery of placenta. (binary)
Breastfeeding within 1 Hour as measured by observer recorded questionnaire | up to 6 months after installation
  Breastfeeding is initiated within one hour of delivery. (binary)
Initial Exam: Previous Pregnancy Inquiry as measured by observer recorded questionnaire | up to 6 months after installation
  Provider asks about complications during previous pregnancies. (binary)
Initial Exam: Hand Washing as measured by observer recorded questionnaire | up to 6 months after installation
  Provider washes his/her hands with soap and water or uses alcohol hand rub before initial examination. (binary)
Initial Exam Temperature Assessment as measured by observer recorded questionnaire | up to 6 months after installation
  Provider takes mother's temperature during initial exam. (binary)
Initial Exam Fundal Height Assessment as measured by observer recorded questionnaire | up to 6 months after installation
  Provider checks fundal height during initial exam. (binary)
Initial Exam Fetal Presentation Assessment as measured by observer recorded questionnaire | up to 6 months after installation
  Provider checks fetal presentation by palpation of abdomen. (binary)
Initial Exam Fetal Heart Rate Assessment as measured by observer recorded questionnaire | up to 6 months after installation
  Provider checks fetal heart rate with fetoscope/Doppler/ultrasound. (binary)
Initial Exam: Vaginal Examination as measured by observer recorded questionnaire | up to 6 months after installation
  Provider performs vaginal examination at initial exam. (binary)
Sterile Gloves for All Exams as measured by observer recorded questionnaire | up to 6 months after installation
  Provider wears sterile gloves for all vaginal examinations. (binary)
Preparation for Delivery: Cord ties/clamps and sterile scissors/blade as measured by observer recorded questionnaire | up to 6 months after installation
  Prepares disposable cord ties/clamps AND sterile scissors/blade. (binary)
Support of Perineum as measured by observer recorded questionnaire | up to 6 months after installation
  Provider supports perineum after baby's head is delivered. (binary)
Cord Traction as measured by observer recorded questionnaire | up to 6 months after installation
  Applies traction to the cord while applying suprapubic counter traction. (binary)
Uterine Massage as measured by observer recorded questionnaire | up to 6 months after installation
  Provider performs uterine massage immediately following the delivery of the placenta. (binary)
Newborn Temperature as measured by observer recorded questionnaire | up to 6 months after installation
  Provider checks newborn's temperature. (binary)
Assistance with Breastfeeding as measured by observer recorded questionnaire | up to 6 months after installation
  Provider assists mother with breastfeeding. (binary)
Sterilization of Equipment as measured by observer recorded questionnaire | up to 6 months after installation
  Provider sterilizes or uses high-level disinfection for all reusable instruments. (binary)
Waste Disposal as measured by observer recorded questionnaire | up to 6 months after installation
  Provider disposes of all contaminated waste in leak-proof containers. (binary)
Hand Hygiene after Clean Up as measured by observer recorded questionnaire | up to 6 months after installation
  Provider washes his/her hands with soap and water or uses alcohol hand rub after cleaning up. (binary)
Delay in Facility Arrival as measured by observer recorded questionnaire | up to 6 months after installation
  Time between facility arrival and first contact with health worker (mins)
Delay in First Exam as measured by observer recorded questionnaire | up to 6 months after installation
  Time between facility arrival and first assessment (mins)
Delay in Uterotonic as measured by observer recorded questionnaire | up to 6 months after installation
  Time between delivery and uterotonic (mins)
Delay in Assessment for Lacerations as measured by observer recorded questionnaire | up to 6 months after installation
  Time between delivery and assessment of perineal and vaginal lacerations (mins)
Delay in Drying Newborn as measured by observer recorded questionnaire | up to 6 months after installation
  Time between delivery and drying baby with towel (mins)
Delay in Breastfeeding Initiation as measured by observer recorded questionnaire | up to 6 months after installation
  Time between delivery and initiation of breastfeeding (mins)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Cohen, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Slawa Rokicki, PhD, Principal Investigator — University College Dublin
Locations (1):
- Innovations for Poverty Action, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
After manuscript publication, fully de-identified data may be shared with researchers upon request.

REFERENCES:
- [Background] Tripathi V, Stanton C, Strobino D, Bartlett L. Development and Validation of an Index to Measure the Quality of Facility-Based Labor and Delivery Care Processes in Sub-Saharan Africa. PLoS One. 2015 Jun 24;10(6):e0129491. doi: 10.1371/journal.pone.0129491. eCollection 2015. PMID 26107655
- [Background] USAID. Maternal and Child Health Integrated Program (MCHIP), Washington DC: USAID/Jhpiego; 2013.
- [Derived] Chang W, Cohen J, Mwesigwa B, Waiswa P, Rokicki S. Impact of reliable light and electricity on job satisfaction among maternity health workers in Uganda: A cluster randomized trial. Hum Resour Health. 2022 Mar 29;20(1):30. doi: 10.1186/s12960-022-00722-3. PMID 35351147
- [Derived] Rokicki S, Mwesigwa B, Schmucker L, Cohen JL. Shedding light on quality of care: a study protocol for a randomized trial evaluating the impact of the Solar Suitcase in rural health facilities on maternal and newborn care quality in Uganda. BMC Pregnancy Childbirth. 2019 Aug 22;19(1):306. doi: 10.1186/s12884-019-2453-x. PMID 31438896

DOCUMENTS (1):
  • Informed Consent Form (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT03589625/ICF_000.pdf